CLINICAL TRIAL: NCT03150875
Title: Efficacy and Safety Evaluation of IBI308 Versus Docetaxel in Patients With Advanced or Metastatic Squamous Cell Lung Cancer After Failure of First-line Platinum-based Therapy- a Randomized, Open-label, Multicenter, Parallel, Phase 3 Study (ORIENT-3)
Brief Title: A Study Comparing the Efficacy and Safety Between IBI308 and Docetaxel in Patients With Advanced or Metastatic NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308C301
Record Dates: First submitted 2017-05-07; First posted 2017-05-12 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBI308 (Experimental): injection; dosage form: 10ml:100mg; frequency: 200mgQ3W; duration: randomization to the date of the first documented tumor progression per RECIST v1.1 criteria
  Interventions: Drug: IBI308
- docetaxel (Active Comparator): injection; dosage form: 1ml:40mg; Frequency: 75mg/m2 Q3W; duration: randomization to the date of the first documented tumor progression per RECIST v1.1 criteria
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: IBI308 — Anti-PD-1 therapy in Chinese squamous NSCLC patients will be investigated in this clinical trial.
  Arms: IBI308
Drug: Docetaxel — As 2nd line treatment to subjects with squamous NSCLC
  Arms: docetaxel

SUMMARY:
Clinical trial results demonstrate that anti-PD-1 antibodies prolonged OS to approximately 9 months compared with 6 months in docetaxel group. Anti-PD-1 therapy in Chinese squamous NSCLC patients will be investigated in this clinical trial.

Additionally, the correlation between PD-L1 expression and the response to IBI308 treatment in Chinese squamous cell NSCLC patients as well as the role of irRECIST in immune checkpoint inhibitor treatment evaluation will also be assessed

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Histologically or cytologically confirmed squamous cell NSCLC
2. Subjects with stage IIIB/stage IV or recurrent disease (not suitable for definitive concurrent chemoradiotherapy) (according to version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) after failure of first-line platinum-based therapy; Subjects who developed recurrent disease <6 months after platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy also could also be eligible.
3. At lease one measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
4. Age ≥ 18 and ≤ 75
5. ECOG performance status 0-1
6. Life expectancy of at least 12 weeks
7. Adequate organ and bone marrow function

   1. CBC: absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; platelet count (PLT) ≥ 100 × 109 / L; hemoglobin content (HGB) ≥ 9.0 g / dL.
   2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; serum albumin ≥ 28 g / L.
   3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance rate (Ccr) ≥ 40 mL / min (calculated using Cockcroft / Gault equation) Female:CrCl= (140-Age) x Weight(kg) x 0.85 72 x Serum creatinine (mg/dL) Male:CrCl= (140-Age) x Weight(kg) x 1.00 72 x Serum creatinine (mg/dL)
8. Subjects of reproductive potential must be willing to use adequate contraception during the course of the study and through 6 months after the last dose of study treatment.
9. Voluntarily signed written informed consent form, willing and able to comply with scheduled visits and other requirements of the study

Exclusion Criteria:

1. EGFR mutation and ALK rearrangement
2. Mixed adeno-squamous carcinoma or other pathological type
3. Prior therapy with anti-PD-1,anti-PD-L1,anti-CTLA4 antibody or docetaxel
4. Have received following treatment:

   1. Received any investigational agent within 4 weeks of the first dose of study treatment.
   2. Received any anti-tumor therapy (chemotherapy, targeted therapy, tumor immunotherapy or arterial embolization) within 3 weeks of the first dose of study treatment.
   3. Received radiotherapy within 4 weeks of the first dose of study treatment.
   4. Received systemic treatment with high-dose corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive drugs within 4 weeks of first dose. Inhaled or topical steroids and adrenal replacement steroid are permitted in the absence of active autoimmune disease.
   5. Received attenuated live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
   6. Received major surgery (such as craniotomy, thoracotomy or laparotomy) within 4 weeks of the first dose of study drugs or open wound, ulcer or fracture.
5. Unrecovered toxicity (grade >1, according to NCI CTCAE 4.03) due to prior anti-tumor therapy before the first dose of study treatment.
6. Subjects with active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis. Subjects with cured childhood asthma, type I diabetes mellitus and hypothyroidism only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
7. Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation
8. Known allergic or hypersensitive to docetaxel, any monoclonal antibody or any other components used in their preparation.
9. Hemoptysis within 4 weeks of randomization (≥ 1/2 spoon per time).
10. Received thoracic radiotherapy >30Gy within 6 months or palliative radiotherapy (brain or bone metastasis) ≤30Gy within 7 days of randomization.
11. Symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis. Subjects should have stable disease more than 4 weeks from first dose of study treatment, with neurological symptoms returned to NCI CTCAE 4.03 grade 0 or 1, are permitted to enroll.
12. Subjects with a history of interstitial lung disease
13. Superior vena caval obstruction syndrome;
14. Uncontrolled third space effusion, eg. ascites or pleural effusion.
15. Uncontrolled concomitant disease, including but not limited to :

    1. Active or poorly controlled severe infection
    2. Human Immunodeficiency Virus (HIV) infection (HIV antibody positive)
    3. Known acute or chronic active hepatitis B (HBV DNA positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection
    4. Active tuberculosis
    5. Symptomatic congestive heart failure (New York Heart Association grade III-IV) or symptomatic, poorly controlled arrhythmia
    6. Uncontrolled hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg)
    7. Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke and transient ischemic attack, within 6 months of enrollment
    8. Concomitant disease needs anticoagulant therapy
    9. Uncontrolled hypercalcemia(Ca2+>1.5mmol/L or Ca >12mg/dl or corrected Serum Calcium >ULN),or Symptomatic hypercalcemia during diphosphonate therapy
    10. Other primary malignancy, with the exception of: (radical Non-melanoma skin cancer or cured cervical in-situ carcinoma;)
16. Subjects with other diseases or abnormal Lab test results which might increase the risk of enrollment and treatment or Interfere with the interpretation of study results could be excluded according to the judgments of investigator.
17. Women who are pregnant or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang
  - Jiangsu Cancer Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Wu L, Yu X, Xing P, Wang Y, Zhou J, Wang A, Shi J, Hu Y, Wang Z, An G, Fang Y, Sun S, Zhou C, Wang C, Ye F, Li X, Wang J, Wang M, Liu Y, Zhao Y, Yuan Y, Feng J, Chen Z, Shi J, Sun T, Wu G, Shu Y, Guo Q, Zhang Y, Song Y, Zhang S, Chen Y, Li W, Niu H, Hu W, Wang L, Huang J, Zhang Y, Cheng Y, Wu Z, Peng B, Sun J, Mancao C, Wang Y, Sun L. Sintilimab versus docetaxel as second-line treatment in advanced or metastatic squamous non-small-cell lung cancer: an open-label, randomized controlled phase 3 trial (ORIENT-3). Cancer Commun (Lond). 2022 Dec;42(12):1314-1330. doi: 10.1002/cac2.12385. Epub 2022 Nov 6. PMID 36336841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Final analysis data cutoff date: 31-July-2020. Of the 290 randomized participants, 14 were ongoing. For efficacy analysis, full analysis set (FAS), Sintilimab (145) and Docetaxel (135), was used. 10 participants in the docetaxel arm who initiated immunotherapy before receving docetaxcel or disease progression were excluded from FAS.
Groups:
- Sintilimab: Sintilimab 200mg Intravenously every 3 weeks
- Docetaxel: Docetaxel 75mg/m2 Intravenously every 3 weeks
Period: Overall Study
Arm/Group | Sintilimab | Docetaxel
Started | 145 | 145
Treated | 144 | 130
Crossover to Certain Treatment | 0 | 0
Completed | 0 | 0
Not Completed | 145 | 145

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sintilimab | Docetaxel | Total
Number analyzed (Participants) | 145 | 135 | 280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (8.19) | 59.5 (8.41) | 60.1 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 136 | 122 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 145 | 135 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 145 | 135 | 280
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 145 | 135 | 280

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death due to any cause.
Time Frame: Through database cutoff date of 31-July-2020 (up to approximately 35 months)
Population: All randomized participants excluding participants in the docetaxel arm who initiated immunotherapy before receiving docetaxel or disease progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab | Docetaxel
Number analyzed (Participants) | 145 | 135
Months | 11.79 [10.28 to 15.27] | 8.25 [6.47 to 9.82]

2. Secondary Outcome: Progression-free Survival by Investigators' Assessment
Description: Progression-free survival (PFS) was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumours (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions, or unequivocal progression of non-target lesion. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS as assessed by investigators per RECIST 1.1 was reported for each arm.
Time Frame: Through database cutoff date of 31-July-2020 (up to approximately 35 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab | Docetaxel
Number analyzed (Participants) | 145 | 135
Months | 4.3 [4.04 to 5.78] | 2.79 [1.91 to 3.19]

3. Secondary Outcome: Overall Response Rate (ORR) Per RECIST v1.1 as Assessed by Investigators
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who experienced a CR or PR is presented.
Time Frame: Through database cutoff date of 31-July-2020 (up to approximately 35 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sintilimab | Docetaxel
Number analyzed (Participants) | 145 | 135
Percentage of participants | 25.5 [18.6 to 33.4] | 2.2 [0.5 to 6.4]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 as Assessed by Investigators
Description: For participants who demonstrated a CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions or unequivoval progression of non-target lesion. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The DOR per RECIST 1.1 for all participants who experienced a CR or PR is presented.
Time Frame: Through database cutoff date of 31-July-2020 (up to approximately 35 months)
Population: All responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab | Docetaxel
Number analyzed (Participants) | 40 | 7
Months | 12.45 [4.86 to 25.33] | 4.14 [1.41 to 7.23]

5. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAE)
Description: TEAE is any AE that developed or worsened in severity compared to the baseline during the period from first dose of any study treatment up to 90 days after the last dose of any study treatment. Percentage of participants experiencing TEAE is calculated.
Time Frame: Through database cutoff date of 31-July-2020 (up to approximately 35 months)
Population: All participants who received ≥1 dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Sintilimab | Docetaxel
Number analyzed (Participants) | 144 | 130
Percentage of participants | 97.20 | 96.20

ADVERSE EVENTS:
Time Frame: Through database cutoff date of 31-July-2020 (up to approximately 35 months)
Description: All adverse events, including serious adverse events, will be collected since the consent form is signed until 90th day after last administration of investigation products, either observed by investigator or by the spontaneous reported by subjects.
Arm/Group | Sintilimab | Docetaxel
All-Cause Mortality (participants affected / at risk) | 108/144 | 101/130
Serious Adverse Events (participants affected / at risk) | 56/144 | 34/130
Other Adverse Events (participants affected / at risk) | 132/144 | 117/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (N=144) | Docetaxel (N=130)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 2
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Myelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 12 | 14
Pneumonia fungal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 4
Platelet count increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Shock (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (N=144) | Docetaxel (N=130)
Anaemia (Blood and lymphatic system disorders) | 48 | 43
Sinus tachycardia (Cardiac disorders) | 12 | 7
Hyperthyroidism (Endocrine disorders) | 11 | 0
Hypothyroidism (Endocrine disorders) | 27 | 2
Constipation (Gastrointestinal disorders) | 23 | 14
Diarrhoea (Gastrointestinal disorders) | 12 | 13
Nausea (Gastrointestinal disorders) | 16 | 12
Vomiting (Gastrointestinal disorders) | 11 | 6
Asthenia (General disorders) | 25 | 33
Chest pain (General disorders) | 8 | 8
Pain (General disorders) | 9 | 3
Pyrexia (General disorders) | 31 | 21
Nasopharyngitis (Infections and infestations) | 9 | 1
Pneumonia (Infections and infestations) | 11 | 11
Upper respiratory tract infection (Infections and infestations) | 17 | 7
Urinary tract infection (Infections and infestations) | 11 | 4
Alanine aminotransferase increased (Investigations) | 25 | 6
Aspartate aminotransferase increased (Investigations) | 23 | 7
Blood bilirubin increased (Investigations) | 9 | 1
Blood urine present (Investigations) | 8 | 1
Gamma-glutamyltransferase increased (Investigations) | 14 | 5
Haemoglobin decreased (Investigations) | 3 | 9
Lymphocyte count decreased (Investigations) | 8 | 9
Neutrophil count decreased (Investigations) | 7 | 38
Platelet count decreased (Investigations) | 6 | 8
Weight decreased (Investigations) | 29 | 14
Weight increased (Investigations) | 10 | 7
White blood cell count decreased (Investigations) | 6 | 39
Decreased appetite (Metabolism and nutrition disorders) | 34 | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 | 13
Hypochloraemia (Metabolism and nutrition disorders) | 13 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 6
Dizziness (Nervous system disorders) | 8 | 3
Headache (Nervous system disorders) | 5 | 7
Proteinuria (Renal and urinary disorders) | 21 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 45
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 0
Rash (Skin and subcutaneous tissue disorders) | 24 | 5
Hypertension (Vascular disorders) | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03150875/Prot_SAP_000.pdf